CLINICAL TRIAL: NCT06961097
Title: The Effect of Virtual Reality Glasess Application on Pain and Anxiety in Women Undergoing Endometrial Biopsy:A Randomized Controlled Research
Brief Title: The Effect of Virtual Reality on Women Undergoing Endometrial Biopsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Sümeyye BAL, Lecturer Ph. D., Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/7/4
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Endometrial Biopsy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): In addition to the routine procedure, virtual reality glasses will be applied to the women in the virtual reality group of the research. After being taken to the gynecological table for the endometraial biopsy procedure, the women included in the experimental group will be made to watch a video lasting an average of 15 minutes with virtual reality glasses until the procedure is completed. While watching the video, the relaxing nature sound music of the video will be played.
  Interventions: Other: Virtual Reality Group
- control group (No Intervention)

INTERVENTIONS:
Other: Virtual Reality Group — control group
  Other Names: control group
  Arms: Virtual Reality Group

SUMMARY:
The aim was to determine the effect of nature sounds and images that will be shown to women who underwent endometrial biopsy by using virtual reality glasses on pain and anxiety.

Hypotheses H0: Virtual reality glasses have no effect on women's pain and anxiety during endometrial biopsy.

H1: Virtual reality glasses have an effect on women's pain and anxiety during endometrial biopsy.

The study will be carried out in two different groups. The practice will start with meeting the women who apply to the Radiology clinic for an endometrial biopsy. After the women are evaluated in terms of eligibility criteria for the research, the women who are eligible will be informed about the research and written informed consent will be obtained from the women who accept. The random distribution of women to the study groups will be carried out using the Block Randomization method. The following applications will be made to the groups.

Virtual Reality Group In addition to the routine procedure, virtual reality glasses will be applied to the women in the virtual reality group of the research. Virtual reality glasses is a device that works on compatible smart mobile phones. After being taken to the gynecological table for the HSG procedure, the women included in the experimental group will be made to watch a video lasting an average of 15 minutes with virtual reality glasses until the procedure is completed. While watching the video, the relaxing nature sounds music of the video will be played in the practice room with a bluetooth speaker.

Control Group Patients in the control group of the study will not be subjected to any treatment other than the routine procedure.

ELIGIBILITY:
Inclusion Criteria:

* *Being over 18 years old

  * Speaking and understanding Turkish
  * Being willing to participate in the research

Exclusion Criteria:

* Not volunteering to participate in research * Not speaking or understanding Turkish

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Scale | immediately before the endometrial biopsy procedure and immediately after the endometrial biopsyprocedure
  It was developed to measure the pain level of patients. It is named differently at two ends on a vertical or horizontal line of ten centimeters (cm) in length (0=no pain, 10=highest level of pain). The numerical values specified by the patient indicate the pain intensity. The validity and reliability of the scale have been performed. It has been determined that it is a suitable method for assessing the pain intensity.
Change in anxiety | immediately before the endometrial biopsy procedure and immediately after the endometrial biopsyprocedure
  STAI-S It is a self-assessment type scale consisting of short statements. While the State Anxiety Inventory (SAI) provides information only about what is felt at that moment, the Trait Anxiety Inventory (TAI) was developed to measure what has been felt in the last 7 days. The SAI-SAI is a Likert-type scale consisting of 20 items and graded from 1 to 4. It is reported that the reliability coefficients obtained as a result of studies conducted with normal and patient samples of the scale vary between .83 and .87

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyye BAL, Ph.D., Study Director — Ondokuz Mayıs University
Locations (1):
- Samsun University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided